CLINICAL TRIAL: NCT05455684
Title: A Randomized, Double-blind, Multicenter, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Aticaprant 10 mg as Adjunctive Therapy in Adult Participants With Major Depressive Disorder (MDD) With Moderate-to-severe Anhedonia and Inadequate Response to Current Antidepressant Therapy
Brief Title: A Study of Aticaprant as Adjunctive Therapy in Adult Participants With Major Depressive Disorder (MDD) With Moderate-to-severe Anhedonia and Inadequate Response to Current Antidepressant Therapy
Acronym: VENTURA-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109217; 67953964MDD3001 (Other: Janssen Research & Development, LLC); 2022-000439-22 (EudraCT Number)
Record Dates: First submitted 2022-07-10; First posted 2022-07-13 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Depressive Disorder, Major; Anhedonia
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia | interventions — Aticaprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aticaprant (Experimental): Participants will receive aticaprant tablets orally once daily for 42 days during double-blind treatment phase in addition to the current antidepressant selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor (SSRI/SNRI) therapy. Participants who will complete the double-blind treatment phase (Day 43) may be eligible to participate in a separate 52-week open-label long-term safety study (67953964MDD3003).
  Interventions: Drug: Aticaprant
- Placebo (Placebo Comparator): Participants will receive matching placebo orally once daily for 42 days during double-blind treatment phase in addition to their current antidepressant (SSRI/SNRI) therapy. Participants who will complete the double-blind treatment phase (Day 43) may be eligible to participate in a separate 52-week open-label long-term safety study (67953964MDD3003).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aticaprant — Aticaprant will be administered orally as tablets.
  Other Names: JNJ-67953964
  Arms: Aticaprant
Other: Placebo — Placebo will be administered orally as tablets.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of aticaprant compared with placebo as adjunctive therapy to an antidepressant in improving depressive symptoms in adult participants with major depressive disorder (MDD) with moderate-to-severe anhedonia (ANH+) who have had an inadequate response to current antidepressant therapy with a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI).

DETAILED DESCRIPTION:
Depression is a common and serious psychiatric disorder which is a leading cause of disability worldwide and is associated with elevated mortality and suicide risk. Aticaprant (JNJ-67953964) is a once daily, highly selective kappa opioid receptor (KOR) antagonist, with demonstrated selectivity over mu opioid receptor (MOR) and delta opioid receptor (DOR) being developed for adjunctive treatment of major depressive disorder (MDD) with moderate-to-severe anhedonia (ANH+). The study consists of a screening phase (up to 30 days prior to randomization), double-blind treatment phase (43 days), and follow-up phase (up to 14 days). The total duration of the study will be up to 87 days. Safety evaluations including adverse events, physical examinations, urine drug test, alcohol breath tests, and clinical laboratory tests will be assessed at specific time points during this study.

ELIGIBILITY:
Inclusion Criteria:

* Be medically stable on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and baseline
* Have a Hamilton Depression Rating Scale 17 item (HDRS-17) total score of 20 or higher at the first and second screening interviews and must not demonstrate a clinically significant improvement between the first and the second independent HDRS-17 assessments
* Meet Diagnostic and Statistical Manual of Mental Disorders-5th edition (DSM-5) diagnostic criteria for recurrent or single episode major depressive disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the structured clinical interview for DSM-5 Axis I disorders-clinical trials version (SCID-CT). Participants 65 years of age or older must have had the first onset of depression prior to 55 years of age
* Have had an inadequate response to at least 1 oral antidepressant treatment, administered at an adequate dose (at or above the minimum therapeutic dose per Massachusetts General Hospital Antidepressant Treatment Response Questionnaire [MGH ATRQ]) and duration (at least 6 weeks) in the current episode of depression. An inadequate response is defined as less than(<) 50% reduction in depressive symptom severity but with some improvement (>0%) (ie, there may be minimal to moderate symptomatic improvement since the initiation of treatment, but some of the initial symptoms are still present, troubling to the participant and affecting behavior and function), as assessed by the MGH ATRQ
* Is currently receiving and tolerating well any one of the following selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) for depressive symptoms at screening, in any approved formulation and available in the participating country/territory: citalopram, duloxetine, escitalopram, fluvoxamine, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, desvenlafaxine at a stable dose for at least 6 weeks. The current antidepressant cannot be the first antidepressant treatment for the first lifetime episode of depression
* Participant's current major depressive episode, and antidepressant treatment response in the current depressive episode, must all be confirmed by the site independent qualification assessment

Exclusion Criteria:

* Have had in the current depressive episode, no response (treatment failure) to 5 or more antidepressant treatments including the current SSRI/SNRI (that is, the one presumed to be continued in the treatment phase) assessed using the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH ATRQ)
* Has a history or evidence of clinically meaningful noncompliance with current antidepressant therapy
* Has a history of moderate-to-severe substance use disorder including alcohol use disorder according to DSM-5 criteria within 6 months before screening
* Has had in the current episode an inadequate response to adequate course of intravenous or intranasal ketamine or esketamine, electroconvulsive therapy, vagal nerve stimulation, or deep brain stimulation device
* Has current, or a history (past 6 months), of seizures
* Has a current homicidal ideation/intent, per the investigator's clinical judgment, or has suicidal ideation with some intent to act within 3 months prior to the start of the Screening Phase, per the investigator's clinical judgment or based on the Columbia Suicide Severity Rating Scale (C-SSRS), corresponding to a response of "Yes" on Item 4 or Item 5, or a history of suicidal behavior within the past 6 months prior to the start of the Screening Phase. Participants reporting suicidal ideation with intent to act or suicidal behavior at baseline should be excluded
* Has one or more of the following diagnoses: a) A DSM-5 diagnosis (which has been the primary focus of psychiatric treatment within the past 2 years) of any of the following: panic disorder, generalized anxiety disorder, social anxiety disorder, specific phobia; b) A current (in the past year) DSM-5 diagnosis of: obsessive-compulsive disorder (OCD), post-traumatic stress disorder (PTSD), anorexia nervosa, bulimia nervosa; c) A current or prior (lifetime) DSM-5 diagnosis of: a psychotic disorder or MDD with psychotic features, bipolar or related disorders, intellectual disability, autism spectrum disorder, borderline personality disorder, antisocial personality disorder, histrionic personality disorder, narcissistic personality disorders, somatoform disorders

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (120):
- United States (46):
  - SW Biomedical Research LLC, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - Advanced Research Center Inc, Anaheim, California
  - Proscience Research Group, Culver City, California
  - Behavioral Research Specialists LLC, Glendale, California
  - Asclepes Research, Long Beach, California
  - Excell Research Inc, Oceanside, California
  - Syrentis Clinical Research, Santa Ana, California
  - Viking Clinical Research Ltd, Temecula, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Innovative Research of West Florida, Incorporated, Clearwater, Florida
  - Vertex Research Group, Inc, Clermont, Florida
  - Gulfcoast Medical Research Center, Fort Myers, Florida
  - New Life Medical Research Center, Inc., Hialeah, Florida
  - Amedica Research Institute Inc, Hialeah, Florida
  - Convenient Medical Center, Hialeah, Florida
  - Galiz Research, Hialeah, Florida
  - Pharmax Research Clinic Inc, Miami, Florida
  - A Plus Research, Miami, Florida
  - Meridian International Research, Miami Gardens, Florida
  - University of Miami, Miami Lakes, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - USF, Department of Psychiatry and Behavioral Neurosciences, Tampa, Florida
  - Research Network America, Berwyn, Illinois
  - Chicago Research Center, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Clinical Trials of America, Monroe, Louisiana
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Psychiatric Care and Research Center (PCRC), O'Fallon, Missouri
  - Bioscience Research LLC, Mount Kisco, New York
  - Fieve Clinical Research Inc, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Montefiore Medical Center PRIME, The Bronx, New York
  - Patient Priority Clinical Sites LLC, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Charak Center for Health and Wellness, Garfield Heights, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - University of Pennsylvania - Perelman School of Medicine, Philadelphia, Pennsylvania
  - West Houston Clinical Research Service, Bellaire, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Bay Area Clinical Services, Friendswood, Texas
  - Clinical Trial Network - Houston, Houston, Texas
  - Alpine Research Organization, Clinton, Utah
  - University of Virginia, Charlottesville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Argentina (8):
  - Hospital Italiano, Buenos Aires
  - STAT Research S A, Buenos Aires
  - CIPREC, Buenos Aires
  - CENydET - Centro Neurobiologico y de Stress Traumatico, Ciudad Autonoma Buenos Aires
  - Fundacion Lennox, Córdoba
  - CENPIA, La Plata
  - Resolution, Mendoza
  - Instituto Medico de La Fundacion Estudios Clinicos, Rosario
- Australia (3):
  - Peninsula Therapeutic & Research Group, Frankston
  - Albert Road Clinic, Melbourne
  - The Alfred Hospital, Melbourne
- Belgium (4):
  - Anima, Alken
  - C.H.U. Brugmann, Brussels
  - Pz Duffel, Duffel
  - Vitaz, Sint-Niklaas
- Brazil (8):
  - Universidade Federal do Ceara Hospital Universitario Walter Cantidio, Fortaleza
  - Instituto Goiano de Neuropsiquiatria, Goiânia
  - NPCRS Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre
  - Ruschel Medicina e Pesquisa Clínica Ltda, Rio de Janeiro
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - CPQuali Pesquisa Clinica LTDA ME, São Paulo
  - BR Trials, São Paulo
- Bulgaria (6):
  - Ambulatory for Individual Practice for Specialized Medical Care in Psychiatry Dr. Ivo Natsov ET, Cherven Bryag
  - Ambulatory Group practice for specialized help in psychiary Philipopolis ODD, Plovdiv
  - Medical Center Mentalcare OOD, Plovdiv
  - Mental Health Center - Rousse, Rousse
  - Medical Center St. Naum, Sofia
  - Mental Health Center - Veliko Tarnovo EOOD, Veliko Tarnovo
- Czechia (7):
  - Narodni ustav dusevniho zdravi, Klecany
  - A Shine S R O, Pilsen
  - Clintrial s r o, Prague
  - AD71 s.r.o., Prague
  - Praglandia s r o, Prague
  - NeuropsychiatrieHK, s.r.o., Prague
  - Psychiatricka ordinace, Ústí nad Labem
- Hungary (7):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Semmelweis Egyetem, Budapest
  - Nyiro Gyula Korhaz, Budapest
  - Bugat Pal Korhaz, Gyöngyös
  - Dr Mathe es Tarsa Bt, Kalocsa
  - PsychoTech Kft, Pécs
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
- Italy (7):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - AUSL LE di Lecce, Lecce
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria alle Scotte, Siena
- Poland (7):
  - Gabinet Lekarski Psychiatryczny Ireneusz Kaczorowski, Bełchatów
  - Mlynowamed Specjalistyczny Psychiatryczny Gabinet Lekarski Joanna Lazarczyk, Bialystok
  - Centrum Badan Klinicznych PI House sp z o o, Gdansk
  - Specjalistyczna Indywidualna Praktyka Lekarska, Lodz
  - SPZOZ Uniwersytecki Szpi.Klin. nr 4 UM w Lodzi, Lodz
  - Osrodek Badan Klinicznych CROMED, Poznan
  - Specjalistyczny Gabinet Psychiatryczny Kowalkowski Gerard, Torun
- Portugal (3):
  - Hospital de Braga, Braga
  - Hospital CUF Inf. Santo, Lisbon
  - Fund. Champalimaud, Lisbon
- Spain (10):
  - Institucion Hosp Hestia Palau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. La Paz, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Univ. Son Espases, Palma de Mallorca
  - Hosp. El Bierzo, Ponferrada
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Alvaro Cunqueiro, Vigo
  - Hosp. Psiquiatrico Alava, Vitoria-Gasteiz
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - ProbarE i Lund AB, Lund
  - ProbarE i Stockholm AB, Stockholm
  - Studieenheten Akademiskt Specialistcentrum Stockholm, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Adult participants aged 18 to 64 years who had major depressive disorder (MDD) with or without moderate-to-severe anhedonia (ANH+ or ANH-) and elderly participants aged 65 to 74 years with MDD (ANH+ and ANH-) who had an inadequate response to an ongoing antidepressant therapy were randomized in the study.
Groups:
- Placebo: During DB treatment phase, participants received placebo matching to aticaprant tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor [SSRI/SNRI]). Participants were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57). Participants who completed the DB phase (at Day 43) and were compliant to the study intervention were eligible to participate in a separate 52-week open-label long-term safety study 67953964MDD3003 (NCT05518149).
- Aticaprant 10 mg: During DB treatment phase, participants received aticaprant 10 mg tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (SSRI/SNRI). Participants were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57). Participants who completed the DB phase (at Day 43) and were compliant to the study intervention were eligible to participate in a separate 52-week open-label long-term safety study 67953964MDD3003 (NCT05518149).
Period: Overall Study
Arm/Group | Placebo | Aticaprant 10 mg
Started | 259 | 254
Safety Analysis Set | 258 | 253
Participants Who Entered Follow-up Phase | 24 | 14
Completed | 244 | 240
Not Completed | 15 | 14
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Adverse Event | 2 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Non-Compliant with study drug | 0 | 1
Not completed — Other | 1 | 2
Not completed — Randomized but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants (adults and elderly) who took at least 1 dose of study intervention.
Groups:
- Placebo: During DB treatment phase, participants received placebo matching to aticaprant tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (SSRI/SNRI). Participants were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57). Participants who completed the DB phase (at Day 43) and were compliant to the study intervention were eligible to participate in a separate 52-week open-label long-term safety study 67953964MDD3003 (NCT05518149).
- Total: Total of all reporting groups
Arm/Group | Placebo | Aticaprant 10 mg | Total
Number analyzed (Participants) | 258 | 253 | 511
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (13.3) | 50.2 (14.6) | 50.8 (13.73)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  Between 18 and 64 years | 213 | 212 | 425
  Between 65 to 74 years | 45 | 41 | 86
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 185 | 184 | 369
  Male | 72 | 69 | 141
  Undifferentiated | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 73 | 71 | 144
  Not Hispanic or Latino | 179 | 176 | 355
  Unknown or Not Reported | 6 | 6 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 5 | 3 | 8
  Black or African American | 25 | 24 | 49
  White | 222 | 213 | 435
  More than one race | 1 | 1 | 2
  Missing or Not reported | 3 | 8 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 18 | 16 | 34
  Australia | 6 | 7 | 13
  Belgium | 12 | 12 | 24
  Brazil | 23 | 18 | 41
  Bulgaria | 17 | 16 | 33
  Czech Republic | 20 | 18 | 38
  Hungary | 2 | 4 | 6
  Italy | 2 | 1 | 3
  Poland | 14 | 17 | 31
  Portugal | 2 | 3 | 5
  Spain | 7 | 9 | 16
  Sweden | 19 | 18 | 37
  United States | 116 | 114 | 230

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 43 in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The scale consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). MADRS total score is the sum of scores from individual question items, which ranges from 0 to 60; higher scores represent a more severe condition. Negative change in MADRS total score indicates improvement.
Time Frame: Baseline (Day 1) to Day 43
Population: Full analysis set (ANH+) included all adult randomized participants with MDD ANH+ who received at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 155 | 158
Units on a scale | -11.4 (0.98) | -12.3 (0.95)
Statistical Analysis 1: Comparison: Placebo vs Aticaprant 10 mg; Test type: Superiority; p = 0.467, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.9, 95% CI 2-sided [-3.24 to 1.49], Standard Error of Mean 1.2

2. Secondary Outcome: Change From Baseline to Day 43 in Dimensional Anhedonia Rating Scale (DARS) Total Score
Description: The DARS is a 17-item self-report questionnaire that is designed to assess anhedonia in MDD across the 4 domains: hobbies, social activities, food/drink, and sensory experience. The DARS scale measures desire, motivation, effort, and consummatory pleasure. The DARS is rated on a 5-point Likert scale (0=not at all, 1=slightly, 2=moderately, 3=mostly, 4=very much) and responses are summed to generate the total score (ranges from 0 to 68). A lower total score is indicative of greater anhedonia. Positive changes in DARS total score indicate improvement.
Time Frame: Baseline (Day 1) to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 139 | 147
Units on a scale | 10.5 (1.50) | 12.0 (1.43)

3. Secondary Outcome: Change From Baseline Over Time in MADRS Total Score
Description: Change from baseline over time in MADRS total score is reported. The MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The scale consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). MADRS total score is the sum of scores from individual question items, which ranges from 0 to 60; higher scores represent a more severe condition. Negative change in MADRS total score indicates improvement.
Time Frame: Baseline (Day 1), Days 15, 29 and 43
Population: Full analysis set (ANH+) included all adult randomized participants with MDD ANH+ who received at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 163 | 166
Units on a scale
  At Day 15 | -5.4 (0.76) | -6.6 (0.72)
  At Day 29: number analyzed (Participants) | 156 | 161
  At Day 29 | -9.4 (0.90) | -11.1 (0.87)
  At Day 43: number analyzed (Participants) | 155 | 158
  At Day 43 | -11.4 (0.98) | -12.3 (0.95)

4. Secondary Outcome: Percentage of Participants Who Achieved Response on Depressive Symptoms Scale Based on MADRS Total Score at Day 43
Description: Percentage of participants who achieved response on depressive symptoms scale based on MADRS total score at Day 43 are reported. Responders are defined as participants with a >=50 percent (%) improvement in the MADRS total score from baseline to a given timepoint. The MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The scale consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). MADRS total score is the sum of scores from individual question items, which ranges from 0 to 60; higher scores represent a more severe condition.
Time Frame: At Day 43
Population: Full analysis set (ANH+) included all adult randomized participants with MDD ANH+ who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 167 | 170
Percentage of participants | 22.8 | 29.4

5. Secondary Outcome: Percentage of Participants With Remission of Depressive Symptoms Based on MADRS Total Score at Day 43
Description: Percentage of participants with remission of depressive symptoms based on MADRS total score at Day 43 is reported. Participant is defined as a remitter at a given time point if the MADRS total score is less than or equal to (<=)10 at that time point. The MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The scale consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). MADRS total score is the sum of scores from individual question items, which ranges from 0 to 60; higher scores represent a more severe condition.
Time Frame: At Day 43
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 167 | 170
Percentage of participants | 12.6 | 17.6

6. Secondary Outcome: Change From Baseline to Day 43 in Patient Health Questionnaire, 9-Item (PHQ-9) Total Score
Description: Change from baseline to Day 43 in PHQ-9 total score is reported. The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) MDD criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 is categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19) and severe (20-27). Negative changes in PHQ-9 total score indicate improvement.
Time Frame: Baseline (Day 1) to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 141 | 149
Units on a scale | -5.9 (0.58) | -6.7 (0.55)
Statistical Analysis 1: Comparison: Placebo vs Aticaprant 10 mg; Test type: Superiority; Least Square Mean Difference = -0.8, 95% CI 2-sided [-2.21 to 0.52], Standard Error of Mean 0.69

7. Secondary Outcome: Change From Baseline Over Time in DARS Total Score
Description: Change from baseline over time in DARS total score is reported. The DARS is a 17-item self-report questionnaire that is designed to assess anhedonia in MDD across the 4 domains: hobbies, social activities, food/drink, and sensory experience. The DARS scale measures desire, motivation, effort, and consummatory pleasure. The DARS is rated on a 5-point Likert scale (0=not at all, 1=slightly, 2=moderately, 3=mostly, 4=very much) and responses are summed to generate the total score (range of 0 to 68). A lower total score is indicative of greater anhedonia. Positive changes in DARS total score indicate improvement.
Time Frame: Baseline (Day 1), Days 15, 29, and 43
Population: Full analysis set (ANH+) included all adult randomized participants with MDD ANH+ who received at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants who were analyzed at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 152 | 147
Units on a scale
  At Day 15: number analyzed (Participants) | 152 | 138
  At Day 15 | 4.8 (1.22) | 5.9 (1.20)
  At Day 29: number analyzed (Participants) | 135 | 139
  At Day 29 | 8.3 (1.38) | 10.0 (1.32)
  At Day 43: number analyzed (Participants) | 139 | 147
  At Day 43 | 10.5 (1.50) | 12.0 (1.43)

8. Secondary Outcome: Change From Baseline Over Time in the PHQ-9 Anhedonia-specific Item (PHQ-9, Item 1)
Description: Change from baseline over time in the PHQ-9 anhedonia-specific item (PHQ-9, item 1 is little interest or pleasure in doing things) is reported. The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) MDD criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 is categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19) and severe (20-27). Negative changes in PHQ-9 total score indicate improvement.
Time Frame: Baseline (Day 1), Day 15, Day 29, and Day 43
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 154 | 149
Units on a scale
  At Day 15: number analyzed (Participants) | 154 | 143
  At Day 15 | -0.4 (1.04) | -0.5 (1.07)
  At Day 29: number analyzed (Participants) | 138 | 143
  At Day 29 | -0.5 (1.04) | -0.8 (1.05)
  At Day 43: number analyzed (Participants) | 141 | 149
  At Day 43 | -0.7 (1.09) | -1.0 (1.09)

9. Secondary Outcome: Percentage of Participants With a Score Less Than (<) 2 in the PHQ-9 Anhedonia-specific Item (PHQ-9, Item 1) at Day 43
Description: Percentage of participants with a score <2 in the PHQ-9 anhedonia-specific item (PHQ-9, item 1 is little interest or pleasure in doing things) at Day 43 is reported. The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) MDD criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 is categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19) and severe (20-27).
Time Frame: At Day 43
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 119 | 128
Percentage of participants | 41.2 | 52.3

10. Secondary Outcome: Change From Baseline Over Time in Patient Reported Outcomes Measurement Information System Short Form - Ability to Participate in Social Roles and Activities - 8a (PROMIS-APS 8a)
Description: Change from baseline over time in the PROMIS-APS 8a is reported. This 8-item measure assesses participants' ability to participate in social roles and activities. The items measures the degree of involvement in social roles, activities, and responsibilities, including work, family, friends, and leisure. Each item is rated on a 5-point ordinal scale including 1=always, 2=usually, 3=sometimes, 4=rarely and 5=never, with higher scores indicating better social functioning. The total scores of PROMIS-APS 8a ranges from 8 to 40 and is transformed using a T-score metric with a mean of 50 and a standard deviation of 10. T-score ranges from 25.9 to 65.4, a higher score indicates better social functioning. Positive change in score indicates improvement.
Time Frame: Baseline (Day 1), Days 15, 29, and 43
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 145 | 150
T-score
  At Day 15 | 2.3 (0.48) | 2.6 (0.46)
  At Day 29: number analyzed (Participants) | 143 | 150
  At Day 29 | 2.8 (0.54) | 3.9 (0.52)
  At Day 43: number analyzed (Participants) | 143 | 148
  At Day 43 | 4.3 (0.63) | 5.5 (0.61)

11. Secondary Outcome: Percent Change From Baseline Over Time in Work Productivity and Activity Impairment: Depression (WPAI:D)
Description: The WPAI:D questionnaire is a validated short instrument that assesses impairment in work and other regular activities over the past 7 days. The WPAI yields four types of scores: (a) Absenteeism (work time missed); (b) Presenteeism (impairment at work / reduced on-the-job effectiveness); (c) Work productivity loss (overall work impairment / absenteeism plus presenteeism); (d) Activity Impairment. The first three scores are derived only for respondents who were working (should be missing for non-working), but the last score is applicable for all respondents. Each score ranges from 0 to 100 with higher scores indicating greater impairment and less productivity. Negative changes in score indicates less impairment and greater productivity.
Time Frame: Baseline (Day 1), Days 29 and 43
Population: Full analysis set (ANH+) included all adult randomized participants with MDD ANH+ who received at least 1 dose of study intervention. As planned overall work impairment (absenteeism plus presenteeism) and activity impairment is reported. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants who were analyzed at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 149 | 154
Percent Change
  Overall work impairment: Day 29: number analyzed (Participants) | 46 | 52
  Overall work impairment: Day 29 | -5.8 (4.59) | -14.2 (4.71)
  Overall work impairment: Day 43: number analyzed (Participants) | 42 | 46
  Overall work impairment: Day 43 | -13.9 (5.07) | -12.9 (5.09)
  Activity impairment: Day29 | -9.2 (2.12) | -13.9 (2.03)
  Activity impairment: Day43: number analyzed (Participants) | 147 | 150
  Activity impairment: Day43 | -13.9 (2.28) | -18.1 (2.20)

12. Secondary Outcome: DB Treatment Phase: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Percentage of participants with TEAEs during DB treatment phase are reported. A TEAE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. A TEAE does not necessarily have a causal relationship with the intervention. TEAEs included both serious and non serious adverse events. TEAEs were defined as AEs with onset during the DB Treatment Phase, or AEs that are a consequence of a pre-existing condition that has worsened since baseline (Day 1).
Time Frame: From start of treatment (Day 1) up to Day 43
Population: Safety analysis set included all randomized participants (adults and elderly) who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Groups:
- DB: Placebo: During DB treatment phase, participants received placebo matching to aticaprant tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (SSRI/SNRI).
- DB: Aticaprant 10 mg: During the DB treatment phase, participants received aticaprant 10 mg tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (SSRI/SNRI).
Arm/Group | DB: Placebo | DB: Aticaprant 10 mg
Number analyzed (Participants) | 258 | 253
Percentage of participants | 39.5 | 45.8

13. Secondary Outcome: Follow-up (FU) Phase: Percentage of Participants With AEs
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Time Frame: From Day 44 up to Day 57
Population: Follow-up analysis set included all randomized participants who entered the follow-up phase after the double-blind treatment phase.
Measure: Number; unit: Percentage of participants
Groups:
- FU: Placebo: Participants who received placebo and completed DB phase entered the follow-up phase and were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57).
- FU: Aticaprant 10 mg: Participants who received aticaprant 10 mg and completed DB phase entered the follow-up phase and were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57).
Arm/Group | FU: Placebo | FU: Aticaprant 10 mg
Number analyzed (Participants) | 24 | 14
Percentage of participants | 8.3 | 7.1

ADVERSE EVENTS:
Time Frame: DB treatment phase: start of treatment (Day 1) up to Day 43, FU Phase: From Day 44 up to Day 57
Description: DB phase: Safety analysis set included all randomized participants (adults and elderly) who received at least 1 dose of study treatment. FU phase population included all randomized participants who entered the FU phase after the double-blind treatment phase.
Groups:
- FU: Placebo: Participants who received placebo and completed DB phase entered follow-up phase and were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57).
- FU: Aticaprant: Participants who received aticaprant 10 mg and completed DB phase entered follow-up phase and were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57).
Arm/Group | DB: Placebo | DB: Aticaprant 10 mg | FU: Placebo | FU: Aticaprant
All-Cause Mortality (participants affected / at risk) | 0/258 | 0/253 | 0/24 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/258 | 3/253 | 0/24 | 0/14
Other Adverse Events (participants affected / at risk) | 34/258 | 54/253 | 0/24 | 1/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=258) | DB: Aticaprant 10 mg (N=253) | FU: Placebo (N=24) | FU: Aticaprant (N=14)
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Suicidal Behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=258) | DB: Aticaprant 10 mg (N=253) | FU: Placebo (N=24) | FU: Aticaprant (N=14)
Diarrhoea (Gastrointestinal disorders) | 8 | 14 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 4 | 0 | 1
Headache (Nervous system disorders) | 22 | 17 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 31 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT05455684/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT05455684/SAP_001.pdf